CLINICAL TRIAL: NCT03310164
Title: The Relationship Between Lung and Gut Microbiome in Chronic Obstructive Pulmonary Disease
Brief Title: Lung and Gut Microbiome in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Bei He, Professor and Chief in Department of Respiratory Medicine, Peking University Third Hospital
Other Study IDs: HB55474
Record Dates: First submitted 2017-10-09; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Throat swab, induced sputum, bronchoalveolar lavage fluid (BALF) and faeces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD: Smokers with clinically stable chronic obstructive pulmonary disease (COPD)
- healthy control: Age-matched subjects without chronic obstructive pulmonary disease (COPD)

SUMMARY:
Increasing evidence have implied that microbiota from airway and gut might be involved in the pathogenesis of chronic obstructive pulmonary disease (COPD). However, the cross-talk between respiratory and gastrointestinal microbiome in COPD is still undetermined. The study is aimed to investigate the interaction between lung and gut flora, and their role in the process of COPD.

DETAILED DESCRIPTION:
Despite the high prevalence of chronic obstructive pulmonary disease (COPD), there continues to be a large gap in our understanding of disease pathogenesis and mechanisms accounting for large variability in disease phenotype. Cigarette smoking is the principal cause of COPD, but only approximately 15% of adults with substantial tobacco exposure develop clinical COPD. Besides, bacterial colonization or infection is also considered as an important factor in COPD. There are very limited data from microbiome studies that suggest that respiratory and gastrointestinal microbiota may be involved in the pathogenesis of COPD. However, the cross-talk between between lung and gut microbiome, and their relationship with various clinical phenotypes of COPD. Here, we conducted 16S rRNA-based pyrosequencing to evaluate the link between the lung-gut axis and the clinical phenotypes of COPD, such as lung function, emphysema, symptoms, exacerbations, inflammation levels and metabolic features.

ELIGIBILITY:
Inclusion Criteria:

1. males aged 40-80;
2. diagnosed with COPD according to the GOLD guidelines;
3. clinically stable patients without medication changes or exacerbation in two months;
4. smoking history of more than 10 pack years

Exclusion Criteria:

1. diagnosed with unstable cardiovascular diseases, significant renal or hepatic dysfunction or mental incompetence;
2. diagnosed with asthma, active pulmonary tuberculosis, diffuse panbronchiolitis, cystic fibrosis, clinically significant bronchiectasis, exacerbation of COPD or pneumonia in two months;
3. prescribed immunosuppressive medications.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinically stable patients with COPD and controls without COPD are enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-06-15 (Actual); Primary Completion 2016-02-15 (Actual); Study Completion 2016-02-15 (Actual)

PRIMARY OUTCOMES:
Microbiota that can predict the progress of lung function | 6 months
  The study is aimed to investigate the relationship between the microbiota and the progress of lung function in COPD

SECONDARY OUTCOMES:
Bacteria related to inflammatory factors | 6 months
  The association between microbiota and inflammatory factors from host is also investigated
Bacteria related to metabolomics | 6 months
  The association between microbiota and metabolites from host is also investigated

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China